CLINICAL TRIAL: NCT03567018
Title: Comprehensive Imaging of Perforator Vessels and Subcutaneous Vascular Network With No-Exogenous Contrast and Non-Ionizing-Radiation Magnetic Resonance Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Wright Center of Innovation in Biomedical Imaging (Unknown)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP0618/2012H0008
Record Dates: First submitted 2018-04-06; First posted 2018-06-25 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Perforator Flap Surgery
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Two populations are being investigated in this trial; a healthy volunteer population and a patient population. Each population will receive an MRI scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Healthy volunteer population (Experimental): We plan to enroll 25 healthy volunteers.
  Interventions: Device: MRI Scan
- Patient population (Experimental): We plan to enroll 50 clinical patients who are receiving flap procedures at the Ohio State Medical Center.
  Interventions: Device: MRI Scan

INTERVENTIONS:
Device: MRI Scan — Study participants will be scanned with a 3.0 Tesla Phillips Ingenia CX whole body clinical MRI system located at the Wright Center of Innovation at The Ohio State University Medical Center. Anatomical and angiographic MR images will be acquired for one of the most commonly used flap surgery donor perforators including but not limited to: the deep inferior epigastric perforators (DIEP); the superior gluteal arter perforators (SGAP); the inferior gluteal artery perforators (IGAP); the thoracodorsal artery perforators (TDAP); the anterolateral thigh perforators (ATL).

SUMMARY:
In this study the investigators plan to enroll a total of 25 evaluable volunteers (volunteer population) for the development and optimization of perforator imaging protocols and 50 evaluable clinical patients receiving flap procedures at OSUMC for the clinical validation of the optimized protocol. No extrinsic MR contrast agent will be injected. Clinical patients' MRI images will be evaluated independently by radiologists and plastic surgeons and compared to the clinical CTA images.

DETAILED DESCRIPTION:
The overall objective of this pilot study is to develop and optimize preoperative MRA imaging protocols for various perforators commonly used in flap surgery with phantoms and healthy volunteers and to obtain clinical validation of the optimized protocols with a group of patients receiving flap surgery at The OSU Wexmer Medical Center. Data obtained in this study may also serve as the basis for statistical planning of future clinical trials. Based on previous experience with other magnetic resonance imaging (MRI) techniques, the investigators hypothesize that optimal MRA images can only be obtained with a carefully selected combination of imaging hardware, acquisition, and postprocessing factors. The main objective of this pilot study is to determine this optimal combination through the comparison of image between different combinations. The secondary objective of this pilot study is to evaluate, both qualitatively and quantitatively, the quality of the optimized MRA images and compare them with clinical CTA images. The primary hypothesis is that the quality of the optimized MRA images is at least comparable to that of the CTA images. The quantitative measurements obtained from this pilot population will also serve as the preliminary data for future studies and be used in statistical calculations that determine their study population.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years at time of enrollment
* able to provide informed consent
* able to lie in both prone and supine positions for at least 30 minutes
* the clinical patients need to have a flap procedure scheduled at the Ohio State University Medical Center within the next 24 months

Exclusion Criteria:

* Use of an IUD (intrauterine device) or medical patch
* Subjects with any type of activatable implants (e.g. cardiac pacemakers, deep brain stimulators, spinal cord stimulators, cochlear implants, electronic infusion pumps, etc.)
* Subjects with any type of metallic implants or foreign objects in torso region (e.g. cardiac stents, surgical clips, shrapnel fragments from war wounds, etc.)
* metal works and machinists (who may have metallic fragments in or near the eyes)
* severe auto accident victims
* subjects with permanent tattoos that may contain metallic coloring
* subjects with previous history of perforator flap surgery
* subjects who cannot communicate with the researcher for any reason
* claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
image quality | through study completion, on average 2-5 years
  assessed by blinded readers
Artifacts in MRI images assessed by experienced readers | through study completion, on average 2-5 years
  assessed by blinded readers
Vessel detectability in MRI assessed by experienced readers | through study completion, on average 2-5 years
  assessed by blinded readers
Image noise as a measure of image quality assessed by quantitative measures | through study completion, on average 2-5 years
  assessed region of interest over target tissue and background

SECONDARY OUTCOMES:
Anatomy accuracy | 60 min
  Location on images
Vascular network continuity | 60 min
  Location on images
Perforator branching pattern | 60 min
  Location on images
Potential Clinical Use of the MRI Images for Clinical Decision making | Baseline
  Clinical reader assessment
Signal-to-noise ratio (SNR) | Baseline
  ROI based assessment
Contrast-to-noise ratio (CNR) to muscle and fat | Baseline
  ROI based assessment
Perforator size | 60 min
  Location on images
Length of perforator intramuscular course | 60 min
  Location on images

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Martha Morehouse Medical Plaza, Columbus, Ohio
  - The Ohio State University Hospital, Columbus, Ohio

DOCUMENTS (1):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT03567018/Prot_000.pdf